CLINICAL TRIAL: NCT05183607
Title: A Cardiac Surgery Virtual Nutrition Intervention Program Feasibility Study-VIP Study
Brief Title: A Cardiac Surgery Virtual Nutrition Intervention Program Feasibility Study-VIP Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Rakesh C. Arora, Section Head and Regional Lead - Cardiac Surgery, St. Boniface Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS25164 (H2021:336)
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Nutritional Deficiency
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Study sessions will be provided using a virtual communication platform and delivered remotely to each participant by a registered dietitian. The virtual counseling sessions will be led by a registered dietitian and delivered to each participant remotely while in the comfort of their own residence or where it is deemed to be comfortable and safe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual nutritional Intervention (Experimental): This arm will receive the virtual nutritional intervention consisting of 4 - 30 minute sessions to educate cardiac surgery patients before their date of surgery. Each session will provide a different theme such as: 1) nutritional assessment, 2) protein intake education, 3) nutritional adequacy prior to surgery, and 4) protein and nutrition intake post surgery
  Interventions: Other: Virtual Nutrition Education

INTERVENTIONS:
Other: Virtual Nutrition Education — 4 interventional sessions will be provided using a virtual communication platform and delivered remotely to each participant by a registered dietitian. The virtual counseling sessions will be led by a registered dietitian and delivered to each participant remotely

SUMMARY:
This feasibility study will look to identify the impact that a remote/virtual nutritional intervention can have on nutrition literacy and knowledge retention of the cardiac surgery patient.

DETAILED DESCRIPTION:
The proposed VIP study will utilize an interventional feasibility design to implement and evaluate the impact of a virtual nutrition intervention prehab program on cardiac surgery patients. The VIP study looks to measure patient adherence and acceptability, and practicality of the remote platform in hopes it will illicit change to the current standard of nutrition care being provided to cardiac surgery patients.

The current standards of care do not call for dietitian involvement for cardiac surgery patients' pre-surgery and little to no involvement for patients not receiving CABG surgery. This feasibility study looks to address this gap in current patient nutrition care.

The study intervention will provide eligible patients (n=20) with access to four 25-30 minute virtual sessions with a registered dietitian during the two-week period prior to surgery. The dietitian will provide the patient with nutrition counseling prior to the patient's elective cardiac surgery. Zoom (or equivalent) software will be utilized as a remote platform to connect the dietitian virtually with participants during all sessions. The four sessions will follow the same presentation format and will provide all participants with identical nutrition education with curriculum content progressing in each subsequent session. Each session will be comprised of protein education and goal setting, with education content building on previous sessions with a goal of improving patient protein intake perioperatively.

Data will be collected on: (1) participant demographics, (2) physical function, (3) nutritional status and (4) nutrition literacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* undergoing non-emergent/elective cardiac surgery

Exclusion Criteria:

* not able to communicate in English (read or write)
* in-patients (urgent or emergent care)
* patients who self report protein supplementation on a regular basis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Nutritional Literacy | Baseline
  measurement of nutrition related understanding - Modified Social Cognitive Theory questionnaire
Nutritional Literacy | 1 week pre-surgery
  measurement of nutrition related understanding - Modified Social Cognitive Theory questionnaire
Nutritional Literacy | I month post Hospital discharge
  measurement of nutrition related understanding - Modified Social Cognitive Theory questionnaire

SECONDARY OUTCOMES:
Nutrition Status - MNA | Baseline
  participant nutritional status - Mini nutritional assessment
Nutrition Status - MNA | 1 week pre-surgery
  participant nutritional status - Mini nutritional assessment
Nutrition Status - MNA | 1 month post Hospital discharge
  participant nutritional status - Mini nutritional assessment
Nutrition Status - BMI | Baseline
  participant nutritional status - Body Mass Index (BMI)
Nutrition Status - BMI | 1 Week pre-surgery
  participant nutritional status - Body Mass Index (BMI)
Nutrition Status - BMI | 1 Month post hospital discharge
  participant nutritional status - Body Mass Index (BMI)
Quality of Life - physical function | Baseline
  modified Short Form - 36 questionnaire to measure physical function
Quality of Life - physical function | 1 week pre-surgery
  modified Short Form - 36 questionnaire to measure physical function
Quality of Life - physical function | 1 month post hospital discharge
  modified Short Form - 36 questionnaire to measure physical function
Nutritional behaviour | Baseline
  3-Day Food Record
Nutritional behaviour | 1 Week pre-surgery
  3-Day Food Record
Nutritional behaviour | 1 month post hospital discharge
  3-Day Food Record
Nutrition Status - PA | Baseline
  participant nutritional status - pre-albumin
Nutrition Status - PA | 1 week pre-surgery
  participant nutritional status - pre-albumin
Nutrition Status - PA | 1 month post hospital discharge
  participant nutritional status - pre-albumin

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Arora, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No